CLINICAL TRIAL: NCT02598024
Title: The Effectiveness of 4-session Narrative Exposure Therapy and 2-session Group Control-focused Behavioural Treatment on PTSD in Nepal Earthquake Survivors After 12 Months: Study Protocol for the Randomised Waiting-list Controlled Trial
Brief Title: Treating Earthquake in Nepal Trauma (TENT) Trial 2016
Acronym: TENT2016
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nepalese Psychological Association (Other)
Responsible Party: Principal Investigator, Suraj Shakya, Clinical Psychologist, Nepalese Psychological Association
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NPA/2/2015
Record Dates: First submitted 2015-10-30; First posted 2015-11-05 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Post-traumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Narrative Exposure Therapy (NET-R) (Experimental): Revised Narrative Exposure Therapy (NET-R) is a 4-session manual-based treatment, each session lasting 60-90-minutes, and first three sessions delivered daily and the last session after a gap of 1-2 days
  Interventions: Behavioral: Narrative Exposure Therapy
- Control Focused Behavioural Treatment (Experimental): CFBT is an intervention to facilitate natural recovery process by restoring sense of control over anxiety, fear, or distress. For this study in Nepal, a monitoring session will be added to the one-session group CFBT used by Basoglu and Salcioglu (2011), and the revised CFBT would be delivered to groups of 20-30 survivors. Each treatment session would be delivered within 1- 2 hours (90 minutes on average), at the interval of two weeks.
  Interventions: Behavioral: Control Focused Behavioural Treatment
- Waiting List Control (No Intervention): The waiting list participants will receive the treatment of choice (NET-R or CBFT-R) after 3 months.

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — In Narrative Exposure Therapy the patient constructs a narration of his or her life, focusing on the detailed context of the traumatic experiences as well as on the important elements of the emotional networks and how they go together. This process allows the majority of persons to recognise that the fear/trauma structure results from past experiences and that its activation is just a memory. They thus lose the emotional response to the recollection of the traumatic events, which consequently leads to a remission of PTSD symptoms. Thus, they gain access to 'lost' past memories and develop a sense of coherence, control, and integration. Revised Narrative Exposure Therapy (NET-R, Zang et al, 2013) is a 4-session treatment delivered within a week.
  Arms: Narrative Exposure Therapy (NET-R)
Behavioral: Control Focused Behavioural Treatment — The Control-focused Behavioural Treatment (CFBT, Başoğlu et al 2005) for earthquake survivors was designed after 1999 Turkey earthquake as an intervention to facilitate natural recovery processes by restoring sense of control over anxiety, fear, or distress. Its underlying principle is to reduce helplessness responses by encouraging behaviours that are likely to enhance sense of control over stressor events and life in general. Its primary aim is to reverse traumatic stress processes by increasing anxiety or distress tolerance. In earthquake survivors, CFBT involves a single session in most cases and an additional few sessions in cases that do not respond to the initial session.
  Arms: Control Focused Behavioural Treatment

SUMMARY:
The purpose of this study is to determine whether two types of short-term trauma-focused therapies (individual Narrative Exposure Therapy and group-based Control-Focused Behavioural Treatment) are effective in the treatment of chronic PTSD in earthquake survivors of Nepal.

DETAILED DESCRIPTION:
Background: Post-traumatic stress disorder (PTSD) is a common mental health disorder after natural disasters. Without treatment survivors of earthquake would continue suffering from PTSD for many years. There are not many short-term trauma-focused psychosocial therapies that have been examined after natural disasters in developing countries. This study investigates the effectiveness of a 4-session revised narrative exposure therapy (NET-R), and 2-session group-based control-focused behavioural treatment (CFBT-R) delivered by non-specialists with minimum supervision.

Methods/Design: Participants would be identified and recruited through a door-to-door survey of families severely affected by the 2015 earthquake in Bhaktpur municipality of Nepal. PTSD Checklist for DSM-5 (PCL-5) will be used to screen all adult survivors (aged 18 and above) for the possible presence of PTSD, and the CAPS-5 interview will be used for the diagnosis of current PTSD. Investigators aim to include 240 consenting participants in a single blind randomised controlled clinical trial. All participants will be randomly allocated to one of three treatment conditions (N = 80 each): 4-session revised narrative exposure therapy (NET-R), 2-session group-based control-focused behavioural treatment (CFBT-R) involving instructions to conduct self-exposure, or a 3-month waiting list. In both NET-R and CFBT-R interventions, treatment sessions will last 90 minutes; NET-R will be delivered within a week while CFBT-R will be done over 2 weeks. All participants will be subjected to blind assessments for PTSD symptom severity with CAPS-5 and Fear and Avoidance questionnaire at pre-treatment (T0) and 3-month post-treatment (T1).

Discussion: The results from the post-treatment measurement would provide strong empirical reference of the safety and effectiveness of trauma-focused short-term therapies (NET-R and CFBT-R) for mass trauma survivors in developing countries like Nepal. It may also provide information on who may benefit most from which type of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Must have a diagnosis of PTSD according to DSM-5 criteria with a Clinically-Administered PTSD Scale (CAPS-5); during the screening, participants will be asked to report on traumatic events that fulfil DSM-5 criterion 'A'.
* The PTSD symptoms must be a result of the Nepal earthquake in April 2015

Exclusion Criteria:

* High suicidality (Yes to the question "Have you recently had thoughts of ending your life and made any plans to this effect?)
* People with severe degree of prolonged grief (Grief Score of 25 or more on the Grief Assessment Scale, adapted from Prigerson et al., 1999)
* Severe intellectual impairment, being unable to communicate and dependent on others for daily living (i.e. suffering from severe Learning disability)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Symptom severity of PTSD as measured by PCL-5 | Pre-treatment (T0), 2-week post-treatment (T1) and at three-month follow-up (T2)
  The PTSD Checklist for DSM-5 (PCL-5; Weathers et al, 2013) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. A total symptom severity score (range - 0-80) can be obtained by summing up the scores for each of the 20 items. The VA National Centre for PTSD has suggested a cut off score of 38 to screen for PTSD.

SECONDARY OUTCOMES:
WHO Disability Assessment Schedule (WHODAS 2) | Pre-treatment (T0), 2-week post-treatment (T1) and at three-month follow-up (T2)
  WHODAS 2 measures disability related to a health condition.
Hopkins Symptom Checklist (HSCL-25) | Pre-treatment (T0), 2-week post-treatment (T1) and at three-month follow-up (T2)
  HSCL is a 25-item instrument to measure depression using DSM-IV criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Arun K Jha, FRCPsych, Study Director — Hertfordshire Partnership University NHS Foundation Trust, UK; Sabitri Sthapit, PhD, Study Chair — Nepalese Psychological Society
Locations (1):
- Nepalese Psychological Association, Ki̇̄rtipur, Kathmandu, Nepal

REFERENCES:
- [Background] Prigerson HG, Shear MK, Jacobs SC, Reynolds CF 3rd, Maciejewski PK, Davidson JR, Rosenheck R, Pilkonis PA, Wortman CB, Williams JB, Widiger TA, Frank E, Kupfer DJ, Zisook S. Consensus criteria for traumatic grief. A preliminary empirical test. Br J Psychiatry. 1999 Jan;174:67-73. doi: 10.1192/bjp.174.1.67. PMID 10211154
- [Result] Basoglu M, Salcioglu E, Livanou M, Kalender D, Acar G. Single-session behavioral treatment of earthquake-related posttraumatic stress disorder: a randomized waiting list controlled trial. J Trauma Stress. 2005 Feb;18(1):1-11. doi: 10.1002/jts.20011. PMID 16281190
- [Result] Zang Y, Hunt N, Cox T. A randomised controlled pilot study: the effectiveness of narrative exposure therapy with adult survivors of the Sichuan earthquake. BMC Psychiatry. 2013 Jan 31;13:41. doi: 10.1186/1471-244X-13-41. PMID 23363689